CLINICAL TRIAL: NCT05843916
Title: Phase III, Open-label, Switch Over Trial of the Efficacy and Safety of Agalsidase Beta Biosidus (AGA BETA BS) in Fabry Disease Patients Previously Stabilized With Fabrazyme®
Brief Title: Switch Over Study of Biosimilar AGA for Fabry Disease
Acronym: SMILE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio Sidus SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-AGA-Fase III-001
Record Dates: First submitted 2022-11-28; First posted 2023-05-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Intervention Model Description: BIO-AGA-Fase III-001 is a Phase III, prospective, multicenter, open-label, single-group, baseline-controlled, switch over clinical trial to evaluate the efficacy and safety of AGA BETA BS in patients with FD already treated and previously stabilized with Fabrazyme®.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGA BETA BS (Experimental): The study has a single-arm. First, all participants will receive 2 doses of Fabrazyme® with approximately 14 days between them, and afterwards all participants will switch treatment and receive AGA BETA BS for 54 weeks
  Interventions: Drug: Recombinant human alpha galactosidase A (agalsidase beta); Drug: Recombinant human alpha-galactosidase A (agalsidase beta)

INTERVENTIONS:
Drug: Recombinant human alpha galactosidase A (agalsidase beta) — All participants will receive 2 doses of Fabrazyme® with approximately 14 days between them. The dose will be 1 mg/kg of body mass every 2 weeks
  Other Names: Fabrazyme
Drug: Recombinant human alpha-galactosidase A (agalsidase beta) — All participants will receive AGA BETA BS for 54 weeks. The dose will be 1 mg/kg of body mass every 2 weeks
  Other Names: AGA BETA BS

SUMMARY:
BIO-AGA-Fase III-001 is a Phase III, prospective, multicenter, open-label, single-group, baseline-controlled, switch over clinical trial to evaluate the efficacy and safety of AGA BETA BS in patients with FD already treated and previously stabilized with Fabrazyme®.

DETAILED DESCRIPTION:
BIO-AGA-Fase III-001 is a Phase III, prospective, multicenter, open-label, single-group, baseline-controlled, switch over clinical trial to evaluate the efficacy and safety of AGA BETA BS in patients with FD already treated and previously stabilized with Fabrazyme®.

The study will be conducted in 2 parts: a 5-week Lead-in period (period 1) and 54 week treatment period (period 2). During period 1 all participants will receive 2 intravenous (IV) infusions of Fabrazyme®, provided by Biosidus. After that, in period 2 all participants will switch treatment to AGA BETA BS.

A total of up to 20 participants are planned for the study.

•The primary objective of the study is to evaluate the equivalence in efficacy between AGA BETA BS and Fabrazyme® after 6 months of treatment in participants with Fabry disease previously stabilized with Fabrazyme, by measuring disease biomarker (mean plasma Lyso-Gb3 marker ratio after 26 weeks of treatment, defined as plasma level of the marker Lyso-Gb3 after 26 weeks (6 months) divided by plasma level of the marker Lyso-Gb3 at baseline).

ELIGIBILITY:
Inclusion Criteria:

Sex and Age

1. Male or female participant with ≥18 and ≤60 years of age at the time of signing the informed consent form (ICF).

   Reproduction
2. Female participants who are not pregnant, breastfeeding, donating eggs (ova, oocytes), or considering becoming pregnant during the study and for 3 months after the last dose of study treatment.
3. All women of childbearing potential (WOCBP) must have a negative urine pregnancy test at the Screening visit and at Baseline visit (prior to the first dose of experimental intervention).
4. WOCBP must use one highly effective form of birth control contraception through the study and for 3 months after the last dose of study treatment (refer to Appendix 1 in Section 10.1).
5. Male participants who are not considering fathering a child during the study and for 3 months after the last dose of study treatment.
6. Male sexually active participant with female partner(s) of childbearing potential must agree to use male condoms during the study and for 3 months after the last dose of study treatment or have documented successful surgical sterilization.

   Informed Consent
7. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

   Type of Participant and Characteristics
8. Confirmed previous diagnosis of FD.

   1. Women: preferably present genetic testing showing pathogenic GLA mutation consistent with FD at screening.
   2. Men: preferably present leukocyte α-Gal A activity below normal range and/ or pathogenic GLA mutation consistent with FD at screening.
   3. At least 50% of the participants will be male with classic FD phenotype. The remaining percentage will consist of male late onset and classic women FD phenotype.
9. Participants who have been on stable Fabrazyme® treatment for at least 6 months prior to Baseline visit.
10. Patients that in the last 3 months before the baseline visit have been receiving ≥80% of Fabrazyme®'s labeled dose/kg, this calculation includes both infusions provided by Biosidus during the Lead in period.
11. Disease status considered clinically stabilized, at Investigators' discretion.
12. Estimated glomerular filtration rate (eGFR) ≥45 mL/minute/1.73 m2 by CKD-EPI equation at Screening visit.
13. If receiving pain killers, angiotensin-converting enzyme (ACE) inhibitors or angiotensin II receptor blockers (ARBs), participants must be in a stable dose for ≥ 4 weeks.

Exclusion Criteria:

Medical Conditions

1. Chronic kidney disease in stage 3b, 4, or 5.
2. History of dialysis, kidney transplant or participants who are on the waiting list for a kidney transplant.
3. Proteinuria ≥1 g/day at screening.
4. Participants who have suffered a clinical cardiovascular event (such as but not limited to myocardial infarction, transient ischemic attack) within 6 months prior to Screening visit.
5. Participants who have clinically significant unstable cardiac disease (such as but not limited to uncontrolled symptomatic arrhythmia, unstable angina, congestive heart failure New York Heart Association class III or IV).
6. Participants who have suffered a clinical cerebrovascular event (such as but not limited to stroke, transient ischemic attack) within 6 months prior to Screening visit.
7. History of anaphylaxis or other type I hypersensitivity reactions to agalsidase beta.
8. History of acute kidney injury in the 12 months prior to Screening visit (such as but not limited to acute interstitial nephritis, acute renal failure of glomerular origin or caused by vasculitis).
9. Presence of any medical, emotional, behavioral, or psychological condition that, according to the Investigator, would interfere with the participant's compliance with the requirements of the study.

   Prior/Concomitant Therapy
10. Treatment initiation or change of dose of ACE inhibitors or ARBs in the 4 weeks before the screening.

    Prior/Concurrent Clinical Trial Experience
11. Current participation in an interventional study, in which the participant received any drug within 90 days before the Screening visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Equivalence in efficacy between AGA BETA BS and Fabrazyme® after 6 months of treatment | 6 months
  • The primary objective of the study is to evaluate the equivalence in efficacy between AGA BETA BS and Fabrazyme® after 6 months of treatment in participants with Fabry disease previously stabilized with Fabrazyme, by measuring disease biomarker. Endpoint: • Mean plasma Lyso-Gb3 marker ratio after 26 weeks of treatment, defined as plasma level of the marker Lyso-Gb3 after 26 weeks (6 months) divided by plasma level of the marker Lyso-Gb3 at baseline.

SECONDARY OUTCOMES:
Difference in efficacy between AGA BETA BS and Fabrazyme® after 1 year of treatment | 1 year
  • To evaluate the difference in efficacy between AGA BETA BS and Fabrazyme® after 1 year of treatment in participants with Fabry disease previously stabilized with Fabrazyme®, by measuring disease biomarker. Endpoint: • Mean plasma Lyso-Gb3 marker ratio after 54 weeks of treatment, defined as plasma level of the marker Lyso-Gb3 after 54 weeks (12 months) divided by plasma level of the marker Lyso-Gb3 at baseline.
Compare the pain severity before and after 26 weeks of treatment with AGA BETA BS | 26 weeks
  • To compare the pain severity before and after the treatment with AGA BETA BS in participants with Fabry disease previously stabilized with Fabrazyme®, as measured by the BPI (Brief Pain Inventory)-short form. Endpoint: • Change from baseline in pain severity as assessed by BPI-short form pain severity items scores after 26 of treatment.
Compare the pain severity before and after 54 weeks of treatment with AGA BETA BS | 54 weeks
  • To compare the pain severity before and after the treatment with AGA BETA BS in participants with Fabry disease previously stabilized with Fabrazyme®, as measured by the BPI (Brief Pain Inventory)-short form. Endpoint: • Change from baseline in pain severity as assessed by BPI-short form pain severity items scores after 54 weeks of treatment.
Compare the impact of pain on daily functions before and after 26 weeks of treatment with AGA BETA | 26 weeks
  • To compare the impact of pain on daily functions before and after the treatment with AGA BETA BS in participants with Fabry disease previously stabilized with Fabrazyme®, as measured by the BPI (Brief Pain Inventory)-short form. Endpoint: • Change from baseline in pain interference as assessed by BPI-short form pain interference items scores after 26 weeks of treatment
Compare the impact of pain on daily functions before and after 54 weeks of treatment with AGA BETA | 54 weeks
  • To compare the impact of pain on daily functions before and after the treatment with AGA BETA BS in participants with Fabry disease previously stabilized with Fabrazyme®, as measured by the BPI (Brief Pain Inventory)-short form. Endpoint: • Change from baseline in pain interference as assessed by BPI-short form pain interference items scores after 54 weeks of treatment
Compare the participants' perception of their own health before and after 26 weeks of treatment with AGA BETA BS | 26 weeks
  • To compare the participants' perception of their own health before and after the treatment with AGA BETA BS in participants with Fabry disease previously stabilized with Fabrazyme®, as measured by the SF (Short Form)-36. Endpoint: • Change from baseline in SF-36 scores after 26 weeks of treatment.
Compare the participants' perception of their own health before and after 54 weeks of treatment with AGA BETA BS | 54 weeks
  • To compare the participants' perception of their own health before and after the treatment with AGA BETA BS in participants with Fabry disease previously stabilized with Fabrazyme®, as measured by the SF (Short Form)-36. Endpoint: • Change from baseline in SF-36 scores after 54 weeks of treatment.
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of platelet count at baseline. | Baseline
  Platelet count at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of platelet count after 14 weeks of treatment. | 14 weeks
  Platelet count at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of platelet count after 26 weeks of treatment. | 26 weeks
  Platelet count at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of platelet count after 54 weeks of treatment. | 54 weeks
  Platelet count at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of red blood cell count at baseline. | Baseline
  Red blood cell count at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of red blood cell count after 14 weeks of treatment | 14 weeks
  Red blood cell count at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of red blood cell count after 26 weeks of treatment | 26 weeks
  Red blood cell count at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of red blood cell count after 54 weeks of treatment | 54 weeks
  Red blood cell count at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hemoglobin at baseline | Baseline
  Hemoglobin at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hemoglobin after 14 weeks of treatment | 14 weeks
  Hemoglobin at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hemoglobin after 26 weeks of treatment | 26 weeks
  Hemoglobin at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hemoglobin after 54 weeks of treatment | 54 weeks
  Hemoglobin at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hematocrit | Baseline
  Hematocrit at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hematocrit | 14 weeks
  Hematocrit at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hematocrit | 26 weeks
  Hematocrit at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of hematocrit | 54 weeks
  Hematocrit at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular volume | Baseline
  Mean corpuscular volume at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular volume | 14 weeks
  Mean corpuscular volume at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular volume | 26 weeks
  Mean corpuscular volume at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular volume | 54 weeks
  Mean corpuscular volume at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular hemoglobin | Baseline
  Mean corpuscular hemoglobin at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular hemoglobin | 14 weeks
  Mean corpuscular hemoglobin at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular hemoglobin | 26 weeks
  Mean corpuscular hemoglobin at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean corpuscular hemoglobin | 54 weeks
  Mean corpuscular hemoglobin at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean cell hemoglobin concentration | Baseline
  Mean cell hemoglobin concentration at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean cell hemoglobin concentration | 14 weeks
  Mean cell hemoglobin concentration at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean cell hemoglobin concentration | 26 weeks
  Mean cell hemoglobin concentration at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of mean cell hemoglobin concentration | 54 weeks
  Mean cell hemoglobin concentration at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of %reticulocytes | Baseline
  %reticulocytes at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of %reticulocytes | 14 weeks
  %reticulocytes at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of %reticulocytes | 26 weeks
  %reticulocytes at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of %reticulocytes | 54 weeks
  %reticulocytes at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of white blood cell count | Baseline
  White blood cell count at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of white blood cell count | 14 weeks
  White blood cell count at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of white blood cell count | 26 weeks
  White blood cell count at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of white blood cell count | 54 weeks
  White blood cell count at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of neutrophils | Baseline
  Neutrophils at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of neutrophils | 14 weeks
  Neutrophils at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of neutrophils | 26 weeks
  Neutrophils at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of neutrophils | 54 weeks
  Neutrophils at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of lymphocytes | Baseline
  Lymphocytes at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of lymphocytes | 14 weeks
  Lymphocytes at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of lymphocytes | 26 weeks
  Lymphocytes at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of lymphocytes | 54 weeks
  Lymphocytes at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of monocytes | Baseline
  Monocytes at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of monocytes | 14 weeks
  Monocytes at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of monocytes | 26 weeks
  Monocytes at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of monocytes | 54 weeks
  Monocytes at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of eosinophils | Baseline
  Eosinophils at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of eosinophils | 14 weeks
  Eosinophils at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of eosinophils | 26 weeks
  Eosinophils at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of eosinophils | 54 weeks
  Eosinophils at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of basophils | Baseline
  Basophils at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of basophils | 14 weeks
  Basophils at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of basophils | 26 weeks
  Basophils at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of basophils | 54 weeks
  Basophils at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of blood urea nitrogen | Baseline
  Blood urea nitrogen at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of blood urea nitrogen | 14 weeks
  Blood urea nitrogen at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of blood urea nitrogen | 26 weeks
  Blood urea nitrogen at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of blood urea nitrogen | 54 weeks
  Blood urea nitrogen at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of phosphate | Baseline
  Phosphate at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of phosphate | 14 weeks
  Phosphate at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of phosphate | 26 weeks
  Phosphate at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of phosphate | 54 weeks
  Phosphate at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of creatinine | Baseline
  Creatinine at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of creatinine | 14 weeks
  Creatinine at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of creatinine | 26 weeks
  Creatinine at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of creatinine | 54 weeks
  Creatinine at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total cholesterol | Baseline
  Total cholesterol at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total cholesterol | 14 weeks
  Total cholesterol at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total cholesterol | 26 weeks
  Total cholesterol at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total cholesterol | 54 weeks
  Total cholesterol at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol LDL | Baseline
  Cholesterol LDL at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol LDL | 14 weeks
  Cholesterol LDL at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol LDL | 26 weeks
  Cholesterol LDL at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol LDL | 54 weeks
  Cholesterol LDL at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol HDL | Baseline
  Cholesterol HDL at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol HDL | 14 weeks
  Cholesterol HDL at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol HDL | 26 weeks
  Cholesterol HDL at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of cholesterol HDL | 54 weeks
  Cholesterol HDL at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of triglycerides | Baseline
  Triglycerides at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of triglycerides | 14 weeks
  Triglycerides at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of triglycerides | 26 weeks
  Triglycerides at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of triglycerides | 54 weeks
  Triglycerides at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of glycemia | Baseline
  Glycemia at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of glycemia | 14 weeks
  Glycemia at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of glycemia | 26 weeks
  Glycemia at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of glycemia | 54 weeks
  Glycemia at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total bilirrubin | Baseline
  Total bilirrubin at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total bilirrubin | 14 weeks
  Total bilirrubin at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total bilirrubin | 26 weeks
  Total bilirrubin at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total bilirrubin | 54 weeks
  Total bilirrubin at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of direct bilirrubin | Baseline
  Direct bilirrubin at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of direct bilirrubin | 14 weeks
  Direct bilirrubin at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of direct bilirrubin | 26 weeks
  Direct bilirrubin at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of direct bilirrubin | 54 weeks
  Direct bilirrubin at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of aspartate aminotransferase | Baseline
  Aspartate aminotransferase at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of aspartate aminotransferase | 14 weeks
  Aspartate aminotransferase at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of aspartate aminotransferase | 26 weeks
  Aspartate aminotransferase at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of aspartate aminotransferase | 54 weeks
  Aspartate aminotransferase at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alanine aminotransferase | Baseline
  Alanine aminotransferase at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alanine aminotransferase | 14 weeks
  Alanine aminotransferase at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alanine aminotransferase | 26 weeks
  Alanine aminotransferase at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alanine aminotransferase | 54 weeks
  Alanine aminotransferase at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of sodium | Baseline
  Sodium at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of sodium | 14 weeks
  Sodium at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of sodium | 26 weeks
  Sodium at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of sodium | 54 weeks
  Sodium at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of potassium | Baseline
  Potassium at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of potassium | 14 weeks
  Potassium at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of potassium | 26 weeks
  Potassium at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of potassium | 54 weeks
  Potassium at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of chlorine | Baseline
  Chlorine at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of chlorine | 14 weeks
  Chlorine at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of chlorine | 26 weeks
  Chlorine at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of chlorine | 54 weeks
  Chlorine at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of bicarbonate | Baseline
  Bicarbonate at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of bicarbonate | 14 weeks
  Bicarbonate at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of bicarbonate | 26 weeks
  Bicarbonate at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of bicarbonate | 54 weeks
  Bicarbonate at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of magnesium | Baseline
  Magnesium at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of magnesium | 14 weeks
  Magnesium at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of magnesium | 26 weeks
  Magnesium at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of magnesium | 54 weeks
  Magnesium at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of calcium | Baseline
  Calcium at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of calcium | 14 weeks
  Calcium at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of calcium | 26 weeks
  Calcium at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of calcium | 54 weeks
  Calcium at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alkaline phosphatase | Baseline
  Alkaline phosphatase at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alkaline phosphatase | 14 weeks
  Alkaline phosphatase at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alkaline phosphatase | 26 weeks
  Alkaline phosphatase at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of alkaline phosphatase | 54 weeks
  Alkaline phosphatase at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total proteins | Baseline
  Total proteins at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total proteins | 14 weeks
  Total proteins at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total proteins | 26 weeks
  Total proteins at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of total proteins | 54 weeks
  Total proteins at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of albumin | Baseline
  Albumin at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of albumin | 14 weeks
  Albumin at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of albumin | 26 weeks
  Albumin at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of albumin | 54 weeks
  Albumin at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of Gamma glutamyl transferase | Baseline
  Gamma glutamyl transferase at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of Gamma glutamyl transferase | 14 weeks
  Gamma glutamyl transferase at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of Gamma glutamyl transferase | 26 weeks
  Gamma glutamyl transferase at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of Gamma glutamyl transferase | 54 weeks
  Gamma glutamyl transferase at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of estimated Glomerular Filtration Rate | Baseline
  estimated Glomerular Filtration Rate at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of estimated Glomerular Filtration Rate | 14 weeks
  estimated Glomerular Filtration Rate at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of estimated Glomerular Filtration Rate | 26 weeks
  estimated Glomerular Filtration Rate at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of estimated Glomerular Filtration Rate | 54 weeks
  estimated Glomerular Filtration Rate at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of urine albumin-creatinine ratio | Baseline
  Urine albumin-creatinine ratio at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of urine albumin-creatinine ratio | 14 weeks
  Urine albumin-creatinine ratio at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of urine albumin-creatinine ratio | 26 weeks
  Urine albumin-creatinine ratio at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of urine albumin-creatinine ratio | 54 weeks
  Urine albumin-creatinine ratio at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the general evaluation of first morning urine | Baseline
  First morning urine at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the general evaluation of first morning urine | 14 weeks
  First morning urine at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the general evaluation of first morning urine | 26 weeks
  First morning urine at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the general evaluation of first morning urine | 54 weeks
  First morning urine at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® regarding cardiac function through the evaluation of electrocardiograms. | Baseline
  General evaluation of cardiac function based on the analysis of electrocardiogram exams performed at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® regarding cardiac function through the evaluation of electrocardiograms. | 26 weeks
  General evaluation of cardiac function based on the analysis of electrocardiogram exam performed after 26 weeks of treatment.
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® regarding cardiac function through the evaluation of electrocardiograms. | 54 weeks
  General evaluation of cardiac function based on the analysis of electrocardiogram exam performed after 54 weeks of treatment.
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® regarding cardiac function through the evaluation of echocardiograms. | Baseline
  Evaluation of cardiac function based on the analysis of bidimensional echocardiogram exam performed at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® regarding cardiac function through the evaluation of echocardiograms. | 26 weeks
  Evaluation of cardiac function based on the analysis of bidimensional echocardiogram exams performed after 26 weeks of treatment.
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® regarding cardiac function through the evaluation of echocardiograms. | 54 weeks
  Evaluation of cardiac function based on the analysis of bidimensional echocardiogram exams performed after 54 weeks of treatment.
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of anti-AGA levels from blood samples. | Baseline
  Evaluation of immunogenicity based on the analysis of anti-AGA levels from blood samples collected at baseline
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of anti-AGA levels from blood samples. | 14 weeks
  Evaluation of immunogenicity based on the analysis of anti-AGA levels from blood samples collected at 14 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of anti-AGA levels from blood samples. | 26 weeks
  Evaluation of immunogenicity based on the analysis of anti-AGA levels from blood samples collected at 26 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the evaluation of anti-AGA levels from blood samples. | 54 weeks
  Evaluation of immunogenicity based on the analysis of anti-AGA levels from blood samples collected at 54 weeks
To characterize the safety of AGA BETA BS treatment in participants with Fabry disease previously stabilized with Fabrazyme® through the analysis of physical assessments, adverse events and infusion-related reactions. | 54 weeks
  Analysis of data obtained from clinical and physical assessments, and from reported adverse events and infusion-related reactions throughout the clinical trial. This outcome will be measured in terms of Presence/Absence of relevant clinical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto A Fernández, MD, Principal Investigator — Instituto de Investigaciones Clínicas Quilmes
Locations (4):
- Argentina (4):
  - Instituto de Nefrología Pergamino S.R.L, Pergamino, Buenos Aires
  - Centro Médico Santa María de la Salud, San Isidro, Buenos Aires
  - Instituto de Investigaciones Clínicas Quilmes, Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba